CLINICAL TRIAL: NCT02642484
Title: Gabapentin in Treatment of Muscle Cramps in Patients With Liver Cirrhosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, Consultant liver and GIT diseases- Tanta university hospital, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sherief Abd-Elsalam
Record Dates: First submitted 2015-12-24; First posted 2015-12-30 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Gabapentin; Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gabapentin (Active Comparator): Gabapentin twice daily
  Interventions: Drug: Gabapentin
- PLacebo (Placebo Comparator): Calcium carbonate twice daily
  Interventions: Drug: Calcium Carbonate

INTERVENTIONS:
Drug: Gabapentin — Gapapentin twice daily
  Other Names: Gaptin
  Arms: Gabapentin
Drug: Calcium Carbonate — calcium carbonate twice daily
  Other Names: Calcitron
  Arms: PLacebo

SUMMARY:
* Muscle cramps markedly affect the quality of life in cirrhotic patients with no highly effective drug.
* Quinine was suggested for treatment of patients with muscle cramps in patients with liver cirrhosis. However, thrombocytopenia, cardiac arrhythmias and cinchonism are serious side effects.

DETAILED DESCRIPTION:
• The aim of the study was to assess the efficacy and safety of Gabapentin in the treatment of muscle cramps in patients with liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* liver cirrhosis patients

Exclusion Criteria:

* allergy to gapabentin.
* pregnancy and lactation. Renal failure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of muscle cramps | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sherief M. Abd-Elsalam, Consultant, Principal Investigator — Hepatology and gastroenterology dept.-Tanta; A. K. Singal, Professor, Principal Investigator — Division of Gastroenterology and Hepatology, UAB, Birmingham, AL, USA; Walaa A. Elkhalawany, Lecturer, Study Director — Hepatology and gastroenterology dept.-Tanta
Locations (1):
- Tanta university - faculty of medicine, Tanta, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided